CLINICAL TRIAL: NCT02111928
Title: NovaTears® Observational Study
Brief Title: NovaTears® Eye Drops Observational Study
Status: Completed | Type: Observational
Sponsor: Novaliq GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: NT-001
Record Dates: First submitted 2014-04-07; First posted 2014-04-11 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NovaTears®
  Interventions: Device: NovaTears® Eye Drops

INTERVENTIONS:
Device: NovaTears® Eye Drops — Topical eye drops for lubrication of the ocular surface

SUMMARY:
This observational pilot-study is intended to collect outcome data from a cohort of 30 patients suffering from hyper-evaporative dry eye disease who are treated with the medical device NovaTears® eye drops for a duration of 5 to 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* According to NovaTears® instruction for use
* ≥ 18 years
* Patients with mild to moderate disease and hyper-evaporative dry eye disease applying eye lid hygiene for at least 14 days
* Ability and willingness to provide written Informed Consent
* Ability and willingness to participate in all examinations
* Willingness and ability to return for follow up visit

Exclusion Criteria:

* Patients with hypersensitivity to any of the components of NovaTears®
* Patients with contact lenses, pregnancies, or who are breast feeding
* Patients with non evaporate dry eye disease
* Patients taking lipid containing eye drops or requiring pharmacologic treatment of dry eye disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mild to moderate hyper-evaporative dry eye disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Efficacy measured by routine ophthalmological assessment | 5 to 7 weeks
  Since this is a naturalistic medical device study under EU legislation, the primary outcome is the performance of the device in the intended indication, i.e. the performance claimed by the manufacturer in the instruction for use as determined by routine ophthalmologic assessments. For NovaTears the performance claimed is lubrication of the eye surface, stabilization of the tear film and relieve of symptoms associated with dry eye. These parameters are operationalized by multiple ophthalmological assessment which are part of routine ophthalmologic examinations including tear fluid volume as determined by the Schirmer I test, stability of the tear film as determined by Tear Film Break-Up Time and relieve of symptoms as determined by subjective patient symptom severity questionnaires and objective assessments of the corneal and conjunctival epithelia.

SECONDARY OUTCOMES:
Local Tolerability measured by ophthalmological assessment | 5 to 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Beckert, MD, Study Director — Novaliq GmbH
Locations (2):
- Germany (2):
  - Zentrum fuer Augenheilkunde Uniklinik Koeln, Cologne
  - Praxis Dr. Kaercher, Heidelberg